CLINICAL TRIAL: NCT01288534
Title: A Study of Hypofractionated Stereotactic Body Radiation Therapy (SBRT) Using Continuous Real-time Evaluation of Prostate Motion
Brief Title: Hypofractionated Stereotactic Body Radiation Therapy (SBRT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Fox Chase Cancer Center (Other); Cedars-Sinai Medical Center (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010.064; HUM00041474 (Other: University of Michigan Medical School IRB)
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Treatment (Experimental)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Patients will receive 5 fractions of radiation (you will not receive radiation therapy on two consecutive days). Each fraction size will be 7.4 Gy. The total dose will be 37 Gy. The 5 treatments will be scheduled to be delivered 2 fractions per business week (Monday through Friday). The total duration of treatment will be no shorter than 15 days and no longer than 19 days.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of using radiation therapy with 5 fractions of radiation to treat prostate cancer with guidance of radiation using the Calypso 4D Treatment System (Calypso).A number of recent studies have used 5 radiation fraction to treat prostate cancer over 2-3 weeks as compared to the typical treatment which would involve 40-42 smaller radiation fractions over 8-9 weeks. This type of radiation using a smaller number of treatments has been called hypofractionated radiation therapy.

The Calypso is a new technique which uses beacons implanted into the prostate which using radio signals are able to localize and track the position of the prostate continuously during radiation therapy. The Calypso system has been approved by the United States Food and Drug Administration (FDA) for guidance of radiation therapy during the treatment of prostate cancer and is being utilized all across the United States. However, it has not been tested for hypofractionated radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed diagnosis of adenocarcinoma of the prostate within 180 days of enrollment
* Signed informed consent
* Gleason score ≤ 7
* If Gleason 7 (3+4=7 or 4+3=7) then <50% of biopsy cores must be positive for any pathologic grade of prostate cancer
* If Gleason score <7 then there is no limit on the percentage of biopsy cores involved by prostate cancer
* PSA (within 90 days prior to enrollment)
* ≤ 15 ng/ml prior to start of therapy if Gleason ≤ 6 and
* ≤ 10 ng/ml prior to start of therapy if Gleason 7
* No plan to use hormone therapy prior to evidence of biochemical failure(ie: No neoadjuvant or adjuvant ADT)
* Tumor stage: T1a, T1b, T1c, T2a, T2b
* ECOG Performance Status 0-1

Exclusion Criteria:

* A history of other malignancy diagnosed within the previous 60 months except for non-melanoma skin cancer.
* Any patients who have received other investigational therapy within the last 60 days
* Individuals that have previously been implanted with permanent Beacon transponders
* Patients that have any prosthetic implants in the pelvic region that contain metal or conductive materials (e.g., an artificial hip)
* Patients with implanted pacemaker or defibrillators
* Patients who are felt to have body habitus not conducive to tracking with Calypso beacons
* Positive lymph nodes or metastatic disease from prostate cancer
* Tumor stage: T2c, T3, or T4
* Previous pelvic radiation therapy
* Previous surgery or chemotherapy for prostate cancer
* Previous transuretheral resection of the prostate (TURP) or cryotherapy to the prostate
* Prior hormone therapy or plans for concurrent or post treatment adjuvant hormonal therapy or chemotherapy
* Hormone therapy to include LHRH agonist or oral anti-androgen
* Finasteride and Dutasteride use not excluded
* Concomitant antineoplastic therapy (including surgery, cryotherapy, conventionally fractionated radiation therapy, and chemotherapy) while on this protocol
* History of Crohn's Disease or Ulcerative Colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Spratt, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - The Radiological Associates of Sacremento, Sacramento, California
  - University of Michigan Cancer Center, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Treatment
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Treatment
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 63 [46 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Minimally Detected Decline (MDD) in Quality of Life (QOL)
Description: To evaluate the safety of the proposed hyperfractionation regimen of 5 fractions of radiation to treat prostate cancer with guidance of radiation using the Calypso 4D Treatment System (Calypso, and to compare it to that expected from conventional treatment, which would involve 40-42 smaller radiation fractions over 8-9 weeks.
  Percentage of patients with a MDD in Quality of Life (QOL) surveys for urinary incontinence (UI), urinary obstructive (UO), bowel (BS), and sexual (SS) domains were reviewed at 6 months and 24 months.
Time Frame: 24 months
Measure: Number; unit: percentage of patients
Arm/Group | Radiation Treatment
Number analyzed (Participants) | 68
percentage of patients
  UI by MDD, 6 Months, n=46 | 17
  UI by MDD, 24 Months, n=34 | 18
  UO by MDD, 6 Months, n=46 | 41
  UO by MDD, 24 Months, n=36 | 19
  BS by MDD, 6 Months, n=45 | 33
  BS by MDD, 24 Months, n=31 | 23
  SS by MDD, 6 Months, n=44 | 39
  SS by MDD, 24 Months, n=35 | 43

2. Secondary Outcome: Percentage of Patients With a PSA Nadir of <3.35 ng/ml at 12 Months
Description: To estimate one year prostate specific antigen (PSA)control of prostate cancer when treated with stereotactic body radiotherapy (SBRT) using continuous real-time evaluation of prostate motion.
Time Frame: 1 Year
Measure: Number; unit: percentage of patients
Arm/Group | Radiation Treatment
Number analyzed (Participants) | 68
percentage of patients | 89

3. Secondary Outcome: Relation Between Dose Distribution and Toxicities.
Description: To look at the relation between dose distribution and toxicities and to determine if reconstructed delivered doses are more predictive of toxicity than planned doses.
Time Frame: 5 years
Population: Data was not collected in full by some centers for their patients and these endpoints couldn't be analyzed.
Arm/Group | Radiation Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Relation Between Reconstructed Delivered Dose Distributions.
Description: To determine the relation between reconstructed delivered dose distributions, accounting for prostate translation and rotation, and tumor control probabilities.
Time Frame: 5 years
Population: Data was not collected in full by some centers for their patients and these endpoints couldn't be analyzed
Arm/Group | Radiation Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Frequency of Required Interventions.
Description: To assess the frequency of required interventions (interruptions) based on real-time prostate translations and rotations to verify that the proposed planning target volume(PTV) margins and action level are appropriate and practical. This will be assessed by the percentage of patients with no interventions for any fraction, the percentage of patients with 1-2 fractions interrupted and the percentage of patients with more than two fractions interrupted and the percentage of patients that had an interruption of the beam at least once for all 5 fractions.
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Radiation Treatment
Number analyzed (Participants) | 68
percentage of participants
  No interruptions for any fraction | 24
  1-2 fractions interrupted | 23
  More than 2 fractions interrupted | 53
  At least 1 interruption for all 5 fractions | 24

ADVERSE EVENTS:
Arm/Group | Radiation Treatment
Serious Adverse Events (participants affected / at risk) | 5/68
Other Adverse Events (participants affected / at risk) | 62/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Treatment (N=68)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 2 (2)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Treatment (N=68)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 24 (28)
Fecal incontinence (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 7 (11)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Proctitis (Gastrointestinal disorders) | 18 (19)
Rectal hemorrhage (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 4 (4)
Renal and urinary disorders - Other (Renal and urinary disorders) | 34 (82)
Urinary frequency (Renal and urinary disorders) | 44 (62)
Urinary incontinence (Renal and urinary disorders) | 9 (10)
Urinary retention (Renal and urinary disorders) | 19 (27)
Urinary tract pain (Renal and urinary disorders) | 8 (9)
Urinary urgency (Renal and urinary disorders) | 34 (51)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (3)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Prostatic pain (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 5 (5)
Testicular pain (Reproductive system and breast disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes